CLINICAL TRIAL: NCT01274000
Title: Phase II Study of YM060 - Double-blind, Parallel-group Comparative Study in Patients (Female) With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: A Study to Evaluate Efficacy of YM060 on Diarrhea-predominant Irritable Bowel Syndrome (D-IBS) in Female Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-CL-701
Record Dates: First submitted 2011-01-05; First posted 2011-01-11 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: diarrhea; IBS; Colonic disease; YM060; Ramosetron
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Colonic Diseases | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo
- YM060 low-dose group (Experimental)
  Interventions: Drug: YM060
- YM060 middle-dose group (Experimental)
  Interventions: Drug: YM060
- YM060 high-dose group (Experimental)
  Interventions: Drug: YM060

INTERVENTIONS:
Drug: YM060 — oral
  Other Names: ramosetron, Irribow
  Arms: YM060 high-dose group; YM060 low-dose group; YM060 middle-dose group
Drug: placebo — oral
  Arms: placebo group

SUMMARY:
A study to verify the superiority of YM060 (ramosetron) to placebo for female patients with diarrhea-predominant irritable bowel syndrome (D-IBS) and to evaluate its safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the Rome III Diagnostic Criteria
* Loose (mushy) or watery stools within the last 3 months
* Abdominal discomfort and/or pain during their non-menstrual period

Exclusion Criteria:

* Patients with a history of surgical resection of the stomach, small intestine or large intestine
* Patients with a history or current diagnosis of inflammatory bowel disease (Crohn's disease or colitis ulcerative)
* Patients with a history or current diagnosis of colitis ischemic
* Patients with a current diagnosis of enteritis infectious
* Patients with a current diagnosis of hyperthyroidism or hypothyroidism
* Patients who are currently participating in another clinical trial (including a post-marketing clinical study) or those who participated in another clinical trial (including a post-marketing clinical study) within 12 weeks before the study
* Patients with a history or current diagnosis of malignant tumor
* Patients with a history of abuse of drugs or alcohol within 1 year or those who are currently abusing them

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 409 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Responder rate of patients reported global assessment of relief of IBS symptoms | for 4 weeks

SECONDARY OUTCOMES:
Responder rate of patients reported assessment of relief of abdominal discomfort and/or pain | for 4 weeks
Responder rate of patients reported assessment of improvement of abnormal bowel habits | for 4 weeks
Change in weekly average scores of stool form (appearance) | Baseline and for 4 weeks
Safety assessed by the incidence of adverse events and abnormal values in lab-tests | for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu

REFERENCES:
- [Derived] Fukudo S, Matsueda K, Haruma K, Ida M, Hayase H, Akiho H, Nakashima Y, Hongo M. Optimal dose of ramosetron in female patients with irritable bowel syndrome with diarrhea: A randomized, placebo-controlled phase II study. Neurogastroenterol Motil. 2017 Jun;29(6). doi: 10.1111/nmo.13023. Epub 2017 Feb 16. PMID 28205278
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=060-CL-701